CLINICAL TRIAL: NCT05489731
Title: Phase I Clinical Study of VIC-1911 Combined With Osimertinib in the Treatment of Advanced Non-small Cell Lung Cancer With EGRF- Mutation
Brief Title: VIC-1911 Combined With Osimertinib for EGFR -Mutant Non-small Cell Lung Cancer
Acronym: VIC-1911
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiesi Yingda Pharmaceutical Technology (Suzhou) Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JSI-1911-102
Record Dates: First submitted 2022-07-29; First posted 2022-08-05 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Advanced Non-small Cell Lung Cancer
MeSH Terms: interventions — osimertinib

STUDY DESIGN:
Intervention Model Description: In the dose escalation phase, a total of 2 groups were planned, and 6-12 patients were expected to be enrolled. In the expansion phase, two cohorts are planned, with each cohort expanding to 20-30 patients, and approximately 40-60 patients are expected to be enrolled. A total of 46 to 72 patients were enrolled in this phase I trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose escalation phase-Dose group 1 VIC-1911 Tablets with Osimertinib Mesylate Tablets (Experimental): Advanced NSCLC patients who experienced first/second-generation EGFR-TKI failure with T790M mutation negative or who experienced third-generation EGFR-TKI failure and a subsequent platinum-based doublet chemotherapy failure
  Interventions: Drug: VIC-1911; Drug: Osimertinib Mesylate Tablets
- Dose escalation stage - Dose group 2 VIC-1911 Tablets with Osimertinib Mesylate Tablets (Experimental): Advanced NSCLC patients who experienced first/second-generation EGFR-TKI failure with T790M mutation negative or who experienced third-generation EGFR-TKI failure and a subsequent platinum-based doublet chemotherapy failure
  Interventions: Drug: VIC-1911; Drug: Osimertinib Mesylate Tablets
- Dose expansion phase VIC-1911 Tablets with Osimertinib Mesylate Tablets (Experimental): Cohort 1: NSCLC patients who experienced first/second-generation EGFR-TKI failure with T790M mutation positive; Cohort 2: NSCLC patients who experienced third-generation EGFR-TKI failure
  Interventions: Drug: VIC-1911; Drug: Osimertinib Mesylate Tablets

INTERVENTIONS:
Drug: VIC-1911 — VIC-1911 tablets for oral administration
Drug: Osimertinib Mesylate Tablets — Osimertinib tablets for oral administration
  Other Names: TAGRISSO

SUMMARY:
This is a nonrandomized, open phase I dose escalation and extension clinical study designed to evaluate Aurora A inhibitor VIC-1911 tablets in combination with oxitinib in Chinese patients with advanced non-small cell lung cancer The safety, tolerability, pharmacokinetic characteristics and preliminary antitumor efficacy were analyzed.

The entire study included the screening period (28 days prior to initialadministration of the investigational drug) and the treatment period (Cycle) EoT is defined as disease progression or intolerable toxicity or premature withdrawal Out]) and the safety follow-up period (28 days after EoT). During dose increments and expansions, subjects followed Safety assessment, PK blood collection, imaging examination and efficacy assessment were performed during the visit plan. Observation subject The safety, tolerability, and occurrence of DLT until disease progression, occurrence of intolerable toxicity, Death, withdrawal of informed consent, loss of follow-up or termination of the study by the sponsor shall prevail.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in clinical research, sign written informed consent, and be able to abide by clinical visits and research Relevant procedures;
2. Male or female patients aged 18-75 (including boundary value) when signing the informed consent form;
3. NSCLC with advanced EGFR mutation positive [exon 19 deletion (19del) and exon 21 L858R (21l858r) point mutation] confirmed by cytology or histology A. only applicable to the dose increasing stage: after receiving the first / second generation EGFR-TKI treatment failure T790M mutation negative or third-generation EGFR-TKI treatment failed, and then received platinum containing dual drug chemotherapy Terminal NSCLC patients after failure; B. only applicable to the expansion phase: (1) queue 1: after the treatment failure of the first / second generation EGFR-TKI NSCLC patients with T790M mutation positive; (2) Cohort 2: NSCLC patients who failed to receive three generations of EGFR-tki treatment;
4. According to RECIST 1.1 standard, patients must have a passing shadow Measurable lesions assessed by imaging examination;
5. The EC0G score is 0 or 1;
6. Estimated survival time ≥ 3 months;
7. Bone marrow reserve and organ function level within 7 days before administration must meet the following requirements:

   1. Bone marrow reserve: hemoglobin (HB) ≥ 9.0 g/dl, absolute neutrophil count （ANC）≥ 1.5 × 109/l, platelet (PLT) ≥ 100 × 109/l, opened during the study treatment period Blood transfusion (whole blood, platelets or red blood cells) is prohibited 1 month before the start;
   2. Coagulation function: international normalized ratio (INR) ≤ 1.5 × Upper normal value (ULN), active Partial prothrombin time (APTT) ≤ 1.5 × ULN；
   3. Liver function: aspartate aminotransferase (AST) and alanine in the absence of liver metastasis Transaminase (ALT) ≤ 2.5 × ULN； In case of liver metastasis, AST and alt ≤ 5.0 × ULN；Total bilirubin in serum (TBIL) ≤ 1.5 × ULN (patients known to have Gilbert syndrome Only when total bilirubin ≤ 3 × ULN, direct bilirubin ≤ 1.5 × In the case of ULN, it will be Consider);
   4. Renal function: creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 40 ml/min (according to Cockcroft-Gault formula);
   5. Cardiac function: left ventricular ejection fraction (LVEF) ≥ 50%; ECG is basically normal,QT interval (QTCF) corrected by fridericia formula: male ≤ 450 ms, female ≤ 470 ms；
8. Qualified patients (male and female) with fertility must agree to give drugs during the trial or at the end of the trial Use reliable contraceptive methods (hormone or barrier method or abstinence) with their partners for at least 6 months Etc.); Women of childbearing age (refer to the appendix of the text for the definition) within 7 days before the first use of the investigational drug The pregnancy test must be negative.

Exclusion criteria：

1. Known allergy to, or hypersensitivity to, VIC-1911, osimertinib, or any of the excipient ingredients
2. Subject has previously discontinued osimertinib due to toxicity or other safety events Interstitial lung disease/non-infectious pneumonia; Symptoms or signs of severe arrhythmia with prolonged QTc interval; Symptomatic congestive heart failure
3. Other side effects caused by previous treatment did not alleviate to CTCAE≤ grade 1, alopecia or otherwise
4. A history of ocular disease was present, and the patient had occlusion of central or branch retinal arteries or veins with visual acuity Significant decline, or a history of visual impairment due to other retinal diseases as determined by an ophthalmologist or Performance
5. The following infectious diseases are known to be active, such as:

   Human immunodeficiency virus antibody (HIV-AB) positive; Hepatitis B surface antigen (HBsAg) positive and HBV-DNA exceeding the upper limit of normal value; Hepatitis C virus antibody (HCV-AB) positive and HCV RNA positive
6. Other active infections requiring intravenous antibiotics within 7 days before administration;
7. Use of potent CYP inducer 28 days before administration or within 5 half-lives of the drug, whichever is longer A guide or inhibitor;
8. Had undergone a major surgical procedure within 28 days prior to drug administration or was expected to require a major procedure during the trial Surgery;
9. Received the latest antitumor therapy (chemotherapy, targeted therapy, radiotherapy, immunotherapy, biological therapy) Therapy or endocrine therapy), less than 5 half-lives after or after the first administration of the drug Less than 28 days (whichever is longer). Had received the drug within 14 days before the first dose with definite resistance The effect of traditional Chinese medicine on tumor;
10. A history of serious cardiovascular and cerebrovascular diseases, including but not limited to:

    uncontrolled hypertension (systolic blood pressure >160 mmHg or shu) after standard clinical treatment Tension >100 mmHg for more than 4 weeks); I have severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias that require clinical intervention, Degree II-III atrioventricular block, etc Patients with grade III-IV cardiac insufficiency according to New York Heart Association (NYHA) criteria Any arterial thromboembolic event, including but not limited to myocardial infarction, occurred within 6 months prior to dosing Plug, transient ischemic attack, unstable angina pectoris or other grade 3 or above cardiovascular and cerebrovascular disease Events; Any factor that increases the risk of prolonged QTc intervals or arrhythmias: e.g., heart failure, hypokalemia Haemaemia, congenital long QT syndrome, or the use of anything known to prolong the QT interval Concomitant drugs (see Appendix of the main text for details), except antibiotics used to prevent or treat infection;
11. Parenchymal or meningeal metastases with clinical symptoms were not eligible for inclusion as judged by the investigator. Such as Previous systemic and radical brain metastases therapy (radiotherapy or surgery) proved stable on imaging It has been maintained for at least 28 days and has stopped systemic hormone therapy for more than 14 days without clinical symptoms Is allowed to enter the group;
12. Suffers from hematological malignancies;
13. Other malignant tumors have been diagnosed within 5 years before the first use of the study drug; Effectively treated skin Basal cell carcinoma, squamous cell carcinoma of the skin, and/or effectively resected cervical cancer in situ and/or breast Except the cancer;
14. Inability to swallow medication;
15. Gastrointestinal diseases that may affect the absorption or tolerability of the trial drug, such as refractory or screening CTCAE> grade 2 gastrointestinal symptoms (e.g., nausea, vomiting, diarrhea, etc.);
16. Patients with difficulty in venous blood collection;
17. Women who have a positive pregnancy test or are breastfeeding during the screening period;
18. Administration of an investigational drug that has undergone clinical trials of other drugs within 28 days prior to administration;
19. Previous treatment with other Aurora kinase inhibitors;
20. Patients with a history of blood donation or blood loss of more than 400 mL 3 months before screening;
21. Anything else that, in the opinion of the investigator, may affect the subject to provide informed consent or follow the protocol Circumstances, or the subject's participation in the trial may affect the results of the trial or their own safety.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2024-02-24 (Estimated); Study Completion 2024-04-24 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (safety and tolerability) | 36 months
  Safety and tolerability assessed by adverse events(AEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Pharmacokinetic PK parameters | C1D1 and C1D4 in the first period
  Cmax
Time to Response | Assessed from the date of the first dose of study drug to the first evidence of disease progression or death, whichever is earlier,Expected to evaluate to 36month
  Length of time from the date of first dose of study drug to the first evidence of objective response (CR,PR)
Disease Control Rate | Assessed from the date of the first dose of study drug to the first evidence of disease progression or death, whichever is earlier,Expected to evaluate to 36month
  Proportion of subjects with best response of CR, PR or stable disease (SD)
Progression-Free Survival | Assessed from the date of the first dose of study drug to the first evidence of disease progression or death, whichever is earlier,Expected to evaluate to 36month
  Length of time from the date of first dose of study drug to the first evidence of disease progression or death, whichever is earlier
Overall Survival | Assessed from the date of the first dose of study drug to the first evidence of disease progression or death, whichever is earlier,Expected to evaluate to 36month
  Length of time from the date of first dose of study drug to date of death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Zhangli, Guangdong, China

IPD SHARING:
Plan to Share IPD: No